CLINICAL TRIAL: NCT03199768
Title: Can the Hospital's Architectural Design Affect the Incidence and Treatment of Delirium in Geriatric Patients? A Comparison Between Single-bed and Multibed Rooms
Brief Title: Delirium in Geriatric Hospital Single-bed and Multibed Rooms
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: Delirium in geriatric patients
Record Dates: First submitted 2017-06-01; First posted 2017-06-27 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2017-10

CONDITIONS: Delirium; Older Patients; Admittance to Single-bed Rooms or Multi-bed Rooms
Keywords: architecture; delirium; environment; hospital design and construction
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single-bed rooms: Patients are admitted to single-bed rooms at the newly built hospital in the period 20th of March to the 1th of September 2017
- Multi-bed rooms: Patients are admitted at multi-bed rooms with one to two fellow patients at the old hospital in the period 15th of September 2016 to the 19th of March 2017

SUMMARY:
To investigate whether single-bed rooms can prevent and reduce incidence and duration of delirium compared to multi-bed rooms in elderly patients admitted to a geriatric department. In addition, it is investigated whether single-bed rooms reduce the use of psychotropic drugs, opioids, parenteral medication, fixed guard, falls, hospitalization and discharge to institution among delirious patients. Furthermore, to study if delirium is associated with of re-hospitalization, traumatic fall, institutionalization and death within 30 days, compared to those who do not develop delirium.

DETAILED DESCRIPTION:
Design:

The project will be conducted as an observational prospective cohort study. Patients hospitalized in the period from the 15th September 2016 to the 1th September 2017 which meet the criteria are included

Inclusion Criteria:

Patients 75 Years and older admitted to Geriatric ward at Aarhus University Hospital.

Exclusion Criteria:

Patients who upon admission are dying assessed by a specialist in geriatrics, Patients with stroke where aphasia is present, Patients with severe dementia without language, Patients who are inability to understand or speak Danish.

Data collection:

All patients who meet the inclusion criteria will be examined for state of delirium by using the Confusion Assessment Method (CAM).

The primary outcome is delirium, diagnosed with positive CAM, which is measured morning and evening every day of the week. Duration of delirium is defined by 1 or more consecutive positive CAM scores, and ends if there have been three consecutive negative CAM scores. During hospitalization, it is registered if the patient is staying in a single or a multi-bed room.

Additionally, it is registered, if the old patient has infections, anemia, hypo-natremia, constipation and urinary retention. In the event of delirium, the consumption of psychiatric drugs and changes in drug administration, need for fixed guard and fall episodes are recorded. In the event of delirium, the consumption of psychiatric drugs and changes in drug administration, need for fixed guard and fall episodes are recorded. Length of hospital stay is calculated and it is recorded if the patients are discharge for home, nursing homes or sheltered housing facilities. Follow-up is 30 days after discharge. Traumatic fall is registered in Emergency Department, housing change, re-hospitalization and death is recorded.

Primary outcome is collected prospectively and secondary outcome is collected retrospectively from the electronic patient journal.

Settings: The daily assessment of delirium is part of the regular procedure in the Geriatric Department.

Halfway through the data collection period, The department of Geriatric moves from old hospital buildings to newly built hospital. At the old hospital there are 2.5% single rooms and at the new 100% single rooms.

Patients are included using civil registration number. They may be hospitalized once at both at the old and the new, but they can not be included twice in the same type of hospital.

Sample size: The power calculation is based on an observation study by Caruso et al. Incidence of delirium in single and multi-beds rooms in intensive patients (mean age 59 years) is compared. The incidence of delirium in single-bed rooms is 6.8% versus 15.1% in multi-bed rooms. With a power of 90% and a significance level of 5%, we need 320 patients in each group (N = 640).

Time frame: On average there are admitted 75 older patients pr. months. We expect that 10% are re-hospitalized. When calculating vacation and re-hospitalization, the data collection period is expected to last 12 months.

ELIGIBILITY:
Inclusion Criteria:

Patients 75 Years and older admitted to Geriatric ward and at Aarhus University Hospital in the period from the 15th of September 2016 to the 1th of September 2017.

Exclusion Criteria:

* Patients who upon admission are dying assessed by a specialist in geriatrics
* Patients with apoplexy where aphasia is present
* Patients with severe dementia without language
* Patients who are inability to understand or speak Danish

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Old patients (aged ≥75 years), acutely admitted to a geriatric ward at Aarhus University Hospital for both diseases that need medical and/or surgical treatment.
Sampling Method: Probability Sample
Enrollment: 1014 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Delirium | Repeated measurements twice a day at 7-11 AM and at 5-10 PM. From first day at admission on the geriatric ward until discharge. The average hospitalization period is 7 days. Longitudinal data collection.
  Delirium diagnosed using the Confusion Assessment Method (CAM) - Danish version. Incidence of delirium is measured by the first positive CAM score. Duration of delirium is defined by 1 or more consecutive positive CAM scores, and ends if there have been three consecutive negative CAM scores. Duration is measured in half days.
Duration of delirium | Repeated measurements twice a day at 7-11 AM and at 5-10 PM. From first day at admission on the geriatric ward until discharge. The average hospitalization period is 7 days. Longitudinal data collection.
  Delirium diagnosed by positive CAM test - Danish version. Incidence of delirium is measured by the first positive CAM score. Duration of delirium is defined by 1 or more consecutive positive CAM scores, and ends if there have been three consecutive negative CAM scores. Duration is measured in half days.

SECONDARY OUTCOMES:
Use of Psychotropic drug | First day at admission on the geriatric ward at 20:00 PM and until discharge. The average length of hospital stay is 7 days.
  By positive CAM: Use of Psychotropic drugs will be recorded from the medical chart.
Changes in medication - Opioid | First day at admission on the geriatric ward at 20:00 PM and until discharge. The average length of hospital stay is 7 days.
  By positive CAM: Changes in opioid will be recorded from the medical chart.
Changes in consumption of medicine | First day at admission on the geriatric ward at 20:00 PM and until discharge. The average length of hospital stay is 7 days.
  By positive CAM: Changes in the consumption of medicine will be recorded from the medical chart.
Fixed guard at the patient | First day at admission on the geriatric ward at 20:00 PM and until discharge. The average length of hospital stay is 7 days.
  By positive CAM: The patient must not be alone in the hospital room. Care staff will be with the patient all the time
Traumatic fall | First day at admission on the geriatric ward at 20:00 PM and until discharge. The average length of hospital stay is 7 days.
  By positive CAM:Traumatic fall under hospitalization will be reported to Danish Patient Safety Authority as an Unintended Event. Retrospective traumatic fall will be recorded
Length of hospital stay (LOS) | First day at admission on the geriatric ward and until discharge. The average length of hospital stay is 7 days.
  Calculated from admission to discharge from the geriatric ward
Discharge to own home or institutionalization | At discharge from geriatric ward. 0-1 hours after discharge.
  Recorded if the patients are discharge for home, nursing homes or sheltered housing facilities. Information will be recorded from the medical chart.
Re-hospitalization | 0-30 days after discharge
  Recorded if the patients are re-hospitalization
Death | 0-365 days after admission
  Date of death within 30, 90 and 365 days after admission

CONTACTS AND LOCATIONS:
Overall Officials: Else Marie Damsgaard, Professor, Study Chair — Department of Geriatrics , Aarhus University Hospital, Palle Juul-Jensens Boulevard 99, Building J, J513, DK-8200 Aarhus N
Locations (1):
- University of Aarhus, Health, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqi N, Harrison JK, Clegg A, Teale EA, Young J, Taylor J, Simpkins SA. Interventions for preventing delirium in hospitalised non-ICU patients. Cochrane Database Syst Rev. 2016 Mar 11;3(3):CD005563. doi: 10.1002/14651858.CD005563.pub3. PMID 26967259
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Result] Caruso P, Guardian L, Tiengo T, Dos Santos LS, Junior PM. ICU architectural design affects the delirium prevalence: a comparison between single-bed and multibed rooms*. Crit Care Med. 2014 Oct;42(10):2204-10. doi: 10.1097/CCM.0000000000000502. PMID 25226117